CLINICAL TRIAL: NCT03691220
Title: Improving Medication Adherence in Adolescents Who Had a Liver Transplant
Acronym: iMALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of California, Los Angeles (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Baylor College of Medicine (Other); University of Pittsburgh (Other); University of California, San Francisco (Other); Children's Hospital of Michigan (Other); Children's Hospital of Philadelphia (Other); Emory-Children's Center (Other); The Hospital for Sick Children (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Columbia University (Other); Seattle Children's Hospital (Other); University of Miami (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Eyal Shemesh, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 18-0061; U01DK119200 (NIH)
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Transplant
Keywords: Intervention; Adherence

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to receive the telemetric intervention or standard of care.
Who Masked: Outcomes Assessor
Masking Description: Study pathologists will perform masked reading of for-cause biopsy slides.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemetric Intervention Arm (Experimental): Adolescent with MLVI>2 to receive the telemetric intervention.
  Interventions: Behavioral: Telemetric Intervention
- Standard of Care Arm (No Intervention): Adolescent with MLVI>2 to receive standard of care.

INTERVENTIONS:
Behavioral: Telemetric Intervention — Calls, scripted by a manual; the frequency of the calls varies with patient's MLVI status and preferences.
  Arms: Telemetric Intervention Arm

SUMMARY:
The study's aim is to test a tailored telemetric intervention to reduce rejection incidence by improving medication adherence in a group of adolescent liver transplant recipients identified as nonadherent by a marker (the Medication Level Variability Index, MLVI).

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized controlled trial. The study will be conducted in transplant centers in the United States and Canada. Estimated final sample size of 140 after attrition. Pediatric adolescent and young adult (age at enrollment ≥12 and < 20) transplant recipients will be eligible for participation in the study. Eligible participants will be randomly assigned to intervention or control group. An interim analysis to evaluate efficacy will be performed. Missing data will not be imputed for secondary analyses.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥ 12 and < 20 years of age at enrollment.
* ≥2.5 years after last liver transplantation.
* Guardian's consent, adolescent assent at enrollment.
* The patient is prescribed tacrolimus.
* The patient's MLVI (SD of tacrolimus) was > 2 when calculated by the site for a period of 2 years prior to the review date

Exclusion Criteria:

* The patient has had transplant of an organ other than liver.
* The patient is currently listed for any organ transplantation.
* The patient is expected to transition to another service (e.g., adult clinic, another
* hospital) during the two years of the study.
* Pregnant patients.
* A temporary exclusion: the patient is not medically stable or was hospitalized for >48 consecutive hours in the past three months.
* Site PI, study PI, or Medical Monitor determines that the patient should not be a candidate for the intervention due to factors that are not covered in the above criteria.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Rejection | 2 Years
  The incidence of biopsy-proven acute cellular rejection (number of patients experiencing at least one episode of rejection) at any time during the 2 years of follow up.Biopsy-confirmed late acute rejection, as determined by the majority of 3 masked readings of liver biopsy images by 3 pathologists that are not from the clinical site at which the patient is treated. Patients with incomplete follow-up (for example due to death, re-transplant, listing for re-transplantation), will be assumed to have experienced a rejection for the purpose of the primary analysis.

SECONDARY OUTCOMES:
The Standard Deviation of A Series Of Tacrolimus Levels (MLVI) | 2 Years
  MLVI = Standard Deviation Of Tacrolimus Blood Levels
Incidence of Locally Determined Biopsy Proven Rejection | 2 Years
Rate Of Locally Determined Biopsy Proven Rejection | 2 Years
Rate of Centrally Determined Biopsy Proven Rejection | 2 Years
Time to Rejection From Enrollment | 2 Years
Occurrence of Death | 2 Years
  Number of deaths
Occurrence of Re-Listing For Transplantation | 2 Years
  Number of participants listing for retransplantation
Mean ALT | 2 Years
  Mean number of achieving above threshold ALT > 150 Alanine Aminotransferase (ALT)
Mean maximal ALT | 2 Years
  mean/maximal and ALT (defined as in MALT as the mean of all levels recorded during the study period and the maximal level recorded during the study period)
Mean gGT | 2 Years
  Mean number of achieving above threshold GGT > 150 Gamma Glutamyl Transferase (gGT)
Mean maximal gGT | 2 Years
  mean/maximal gGT (defined as in MALT as the mean of all levels recorded during the study period and the maximal level recorded during the study period)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shemesh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (13):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Benioff Children's Hospital UCSF, San Francisco, California
  - Miami Transplant Institute, Miami, Florida
  - Children's Healthcare of Atlanta/Emory, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - C.S.Mott Children's Hospital, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
- The Hospital For Sick Children Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- See also: Official Website of The iMALT Study — https://imalt.org/